CLINICAL TRIAL: NCT04619966
Title: Ultrasound Measurements of Hepatic Vasculatures and Hepatic Doppler Assessment of Healthy Children
Status: Recruiting | Type: Observational
Sponsor: Hong Kong Children's Hospital (Other)
Responsible Party: Principal Investigator, Pui Kwan Joyce Chan, Associate consultant radiologist, Deputy Head of Ultrasound team of radiology, Principle investigator, Hong Kong Children's Hospital
Other Study IDs: HKCHUSG01
Record Dates: First submitted 2020-10-29; First posted 2020-11-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Portal Vein; Hepatic Veins; Hepatic Artery; Liver Circulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Flow dynamics in the liver is altered in different hepatobiliary and cardiac pathologies, causing changes in hepatic vasculatures sizes and flow pattern changes which can be assessed by ultrasound (USG) study. Before one can use these measurements and observations to diagnose pathologies, a clear grasp of normality is crucial.

In the field of pediatrics, this is particularly challenging as the normal range of measurements may change with age, weight, height, gender and race of children.

Taking hepatic veno-occlusive disease as an example, current literature is conflicting regarding whether sonographic findings show consistent association with the disease. Sonographic findings therefore now have limited role in contributing to the diagnosis.

This may be related to the lack of a robust age corrected normal range of measurement for reference.

Existing literature shows that the normal portal vein diameter varies with age, weight and height and possibly gender. Literature for normal measurements of hepatic vein and hepatic artery in children is lacking.

In this study, the investigators aim to conduct a prospective, cross-section observational study to establish the normal measurements ranges of hepatic vein, hepatic artery and portal vein in healthy children in the investigators' locality.

Flow patterns, including qualitative assessment and quantitative measurements of resistive index and flow velocities will also be assessed.

These age corrected normal measurements will be very helpful in the diagnosis and follow-up of hepatobiliary and cardiac pathologies associated with alterations in dynamics of hepatic circulation.

DETAILED DESCRIPTION:
Trial Objectives and Purpose:

1. To establish normal limits of diameter of hepatic vein, hepatic artery and portal vein according to age, weight, height and gender.
2. To establish normal waveform pattern in ultrasound Doppler assessment of hepatic vein, hepatic artery and portal vein. (Qualitative analysis)
3. To establish normal limits of flow parameters assessed by ultrasound Doppler in hepatic vein, hepatic artery and portal vein according to age, weight, height and gender.

Trial Design:

A prospective cross-section observational study.

Recruitment of study subjects:

Patients attending Hong Kong Children's Hospital for clinically indicated USG examination will be invited to participate in this study under specific inclusion and exclusion criteria.

Treatment of subjects:

Recruited subjects will proceed to the clinically indicated USG study they are referred for first. After the clinically indicated USG study is completed, additional USG & Doppler assessment of hepatic vasculatures will be performed, taking an additional 5 - 10 minutes.

All examinations will be done using a Philips EPIQ 5G ultrasound machine. Curvilinear or linear probe will be used depending on subjects' physique. Size measurements, qualitative and quantitative Doppler assessment of hepatic vein, hepatic artery and portal vein will be made and recorded.

Statistical method to be employed:

Continuous variables will be tested for normality by Shapiro-Wilk's test. Simple statistics including mean and standard deviations (+/- 2 SD) will be used to determine normal ranges for age.

Comparisons will be done by student's t-test. Relations between height, weight and gender with vessels diameter will be tested by Pearson correlation.

Linear multiple regression analysis will be utilized with vessels diameter as the dependent variable.

Number of subject to be enrolled (observation study): 300

Rationale:

Sample size = (Standard normal variate)2 X (Standard deviation)2 / Presicion2 Sample size = 1.962 X 22 / 12 Sample size = 15.37

Standard normal variate = 1.96 at 5% Type I error Standard deviation = up to 2mm (from prior study of portal vein diameter) Precision = 1mm

In view of aim of determining age corrected normal range of vessels diameter in children, a much bigger sample size will be obtained to improve accuracy.

Target to include 300 children in this study.

Age groups:

Around 30 cases for each of the following age groups:

1. 0 - 1 years old
2. 1 - 2 years old
3. 2 - 4 years old
4. 4 - 6 years old
5. 6 - 8 years old
6. 8 - 10 years old
7. 10 - 12 years old
8. 12 - 14 years old
9. 14 - 16 years old
10. 16- 18 years old

ELIGIBILITY:
Inclusion Criteria:

1. Patient < / = 18 years of age.
2. No history of hepatobiliary nor cardiac pathology as checked with record in ePR. Verbal confirmation will be done with patient or parent / legal guardian.
3. Attending USG study other than that of the hepatobiliary system. (ie. Patients attending for thyroid USG, urinary system USG, musculoskeletal system USG etc.)

Exclusion Criteria:

1. Patient > 18 years of age
2. Known history of hepatobiliary or cardiac pathology.
3. Unstable patients.
4. Intolerance of USG examination
5. Uncooperative patients.
6. Patient requiring sedation for USG study.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients attending Hong Kong Children's Hospital for clinically indicated USG examination will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hepatic veins diameter (in mm) measured by grey scale ultrasound at 1 - 2 cm from confluence with inferior vena cava | Baseline
  Right, middle and left hepatic vein diameter (in mm) measured by grey scale Ultrasound at location 1 - 2 cm from confluence with inferior vena cava, measured in longitudinal axis
Hepatic veins Doppler assessment of flow direction (towards or away from inferior vena cava) | Baseline
  Ultrasound Doppler assessment of right, middle and left hepatic veins for flow direction (towards or away from inferior vena cava)
Hepatic veins Doppler assessment of flow pulsatility (yes or no) | Baseline
  Ultrasound Doppler assessment of right, middle and left hepatic veins for flow pulsatility (yes or no)
Hepatic veins Doppler assessment of flow phasicity (monophasic, biphasic or triphasic) | Baseline
  Ultrasound Doppler assessment of right, middle and left hepatic veins for flow phasicity (monophasic, biphasic or triphasic)
Hepatic veins Quantitative Doppler measurement of maximum flow rate (cm/s) | Baseline
  Ultrasound Doppler quantitative measurement of right, middle and left hepatic veins maximum flow rate (cm/s)
Hepatic veins Quantitative Doppler measurement of minimum flow rate (cm/s) | Baseline
  Ultrasound Doppler quantitative measurement of right, middle and left hepatic veins minimum flow rate (cm/s)
Hepatic veins Quantitative Doppler measurement of pulsatility index (only if pulsatility is present) | Baseline
  Ultrasound Doppler quantitative measurement of right, middle and left hepatic veins pulsatility index (Only if pulsatility is present)
Hepatic artery diameter (in mm) measured by grey scale ultrasound at liver hilum | Baseline
  Hepatic artery diameter (in mm) measured by grey scale ultrasound at the hepatic hilum (longitudinal axis)
Hepatic artery Doppler assessment of flow direction (hepatofugal or hepatopetal) | Baseline
  Ultrasound Doppler assessment of hepatic artery flow direction (hepatofugal or hepatopetal)
Hepatic artery Doppler assessment of flow pulsatility (yes or no) | Baseline
  Ultrasound Doppler assessment of hepatic artery flow pulsatility (yes or no)
Hepatic artery Doppler assessment of flow phasicity (monophasic, biphasic or triphasic) | Baseline
  Ultrasound Doppler assessment of hepatic artery flow phasicity (monophasic, biphasic or triphasic)
Hepatic artery quantitative Doppler measurement of peak systolic velocity (cm/s) | Baseline
  Ultrasound Doppler quantitative measurement of hepatic artery peak systolic velocity (cm/s)
Hepatic artery quantitative Doppler measurement of end diastolic velocity (cm/s) | Baseline
  Ultrasound Doppler quantitative measurement of hepatic artery end diastolic velocity (cm/s)
Hepatic artery quantitative Doppler measurement of pulsatility index | Baseline
  Ultrasound Doppler quantitative measurement of hepatic artery pulsatility index
Hepatic artery quantitative Doppler measurement of resistive index | Baseline
  Ultrasound Doppler quantitative measurement of hepatic artery resistive index
Hepatic artery quantitative Doppler measurement of flow volume (ml/s) (measured if feasible) | Baseline
  Ultrasound Doppler quantitative measurement of hepatic artery flow volume (ml/s)
Portal vein diameter (in mm) measured by grey scale ultrasound at liver hilum | Baseline
  Portal vein diameter (in mm) measured by grey scale ultrasound at liver hilum (longitudinal axis)
Portal vein Doppler assessment of flow direction (hepatopetal or hepatofugal) | Baseline
  Ultrasound Doppler assessment of portal vein flow direction (hepatopetal or hepatofugal)
Portal vein Doppler assessment of flow pulsatility (yes or no) | Baseline
  Ultrasound Doppler assessment of portal vein pulsatility (yes or no)
Portal vein Doppler assessment of flow phasicity (monophasic, biphasic or triphasic) | Baseline
  Ultrasound Doppler assessment of portal vein flow phasicity (monophasic, biphasic or triphasic)
Portal vein quantitative Doppler measurement of maximum flow rate (cm/s) | Baseline
  Ultrasound Doppler quantitative measurement of portal vein maximum flow rate (cm/s)
Portal vein quantitative Doppler measurement of minimum flow rate (cm/s) | Baseline
  Ultrasound Doppler measurement of portal vein minimum flow rate (cm/s)
Portal vein quantitative Doppler measurement of pulsatility index (only if pulsatility is present) | Baseline
  Ultrasound Doppler quantitative measurement of portal vein pulsatility index
Portal vein quantitative Doppler measurement of flow volume (ml/s) | Baseline
  Ultrasound Doppler measurement of portal vein flow volume (ml/s)

CONTACTS AND LOCATIONS:
Overall Officials: Pui Kwan Joyce Chan, MBChB, Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patriquin HB, Perreault G, Grignon A, Boisvert J, Filiatrault D, Garel L, Blanchard H. Normal portal venous diameter in children. Pediatr Radiol. 1990;20(6):451-3. doi: 10.1007/BF02075206. PMID 2392362
- [Background] Soyupak S, Gunesli A, Seydaoglu G, Binokay F, Celiktas M, Inal M. Portal venous diameter in children: normal limits according to age, weight and height. Eur J Radiol. 2010 Aug;75(2):245-7. doi: 10.1016/j.ejrad.2009.03.052. Epub 2009 May 5. PMID 19409745
- [Background] Weinreb J, Kumari S, Phillips G, Pochaczevsky R. Portal vein measurements by real-time sonography. AJR Am J Roentgenol. 1982 Sep;139(3):497-9. doi: 10.2214/ajr.139.3.497. No abstract available. PMID 6981312
- [Background] Jequier S, Jequier JC, Hanquinet S, Gong J, Le Coultre C, Belli DC. Doppler waveform of hepatic veins in healthy children. AJR Am J Roentgenol. 2000 Jul;175(1):85-90. doi: 10.2214/ajr.175.1.1750085. PMID 10882252
- [Background] Herbetko J, Grigg AP, Buckley AR, Phillips GL. Venoocclusive liver disease after bone marrow transplantation: findings at duplex sonography. AJR Am J Roentgenol. 1992 May;158(5):1001-5. doi: 10.2214/ajr.158.5.1566656.
- [Background] McCarville MB, Hoffer FA, Howard SC, Goloubeva O, Kauffman WM. Hepatic veno-occlusive disease in children undergoing bone-marrow transplantation: usefulness of sonographic findings. Pediatr Radiol. 2001 Feb;31(2):102-5. doi: 10.1007/s002470000373. PMID 11214676
- [Background] Hommeyer SC, Teefey SA, Jacobson AF, Higano CS, Bianco JA, Colacurcio CJ, McDonald GB. Venocclusive disease of the liver: prospective study of US evaluation. Radiology. 1992 Sep;184(3):683-6. doi: 10.1148/radiology.184.3.1509050.
- [Background] Corbacioglu S, Carreras E, Ansari M, Balduzzi A, Cesaro S, Dalle JH, Dignan F, Gibson B, Guengoer T, Gruhn B, Lankester A, Locatelli F, Pagliuca A, Peters C, Richardson PG, Schulz AS, Sedlacek P, Stein J, Sykora KW, Toporski J, Trigoso E, Vetteranta K, Wachowiak J, Wallhult E, Wynn R, Yaniv I, Yesilipek A, Mohty M, Bader P. Diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in pediatric patients: a new classification from the European society for blood and marrow transplantation. Bone Marrow Transplant. 2018 Feb;53(2):138-145. doi: 10.1038/bmt.2017.161. Epub 2017 Jul 31. PMID 28759025